CLINICAL TRIAL: NCT03664089
Title: Physical Activity Intervention for Gestational Diabetes
Acronym: GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Keim (Other)
Collaborators: Ohio Department of Health (Unknown); Ohio State University (Other); American Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Sarah Keim, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-00178
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Women will receive the standard recommendation for engaging in 150 minutes of physical activity per week, ankle weights (2.5 pounds [1.1 kg]/ankle), instructions on ankle weight usage (wear during normal activity for 2 hours/day, 7 days/week). The weight type and weight amount were chosen based on previously published literature and used in our preliminary work.
  Interventions: Behavioral: Ankle weights (2.5 pounds [1.1 kg]/ankle)
- Control (Placebo Comparator): All women in the control group will receive the standard recommendation for engaging in 150 minutes of physical activity per week.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Ankle weights (2.5 pounds [1.1 kg]/ankle) — Women will receive the standard recommendation for engaging in 150 minutes of physical activity per week, ankle weights (2.5 pounds [1.1 kg]/ankle), documentation for ankle weight usage, an accelerometer, and instructions for accelerometer usage.
  Arms: Intervention
Behavioral: Control — Women will receive the standard recommendation for engaging in 150 minutes of physical activity per week.
  Arms: Control

SUMMARY:
Gestational diabetes mellitus (GDM) portends an immediate, increased risk for Type 2 diabetes mellitus (T2DM). The increased risk associated with having GDM is compounded by excess weight retention. Therefore, the weeks and months immediately after a GDM-complicated pregnancy present an optimal window to initiate lifestyle changes to prevent or delay T2DM. The long-term goal is to prevent T2DM among women with GDM. This study's objective is to evaluate the efficacy of a novel, yet simple, activity-boosting intervention on weight loss among women with GDM.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) portends an immediate, increased risk for Type 2 diabetes mellitus (T2DM). The increased risk associated with having GDM is compounded by excess weight retention, a common issue after any pregnancy. Considering excess weight is the best predictor of developing T2DM, the weeks and months immediately after a GDM-complicated pregnancy present an optimal window to initiate lifestyle changes to prevent or delay T2DM. The long-term goal is to prevent T2DM among women with GDM. This study's objective is to evaluate the efficacy of a novel, yet simple, activity-boosting intervention on weight loss among women with GDM in a parallel two-arm randomized controlled trial (n=80 women/arm, N=160). The intervention uses ankle weights (2.5 pounds [1.1 kg]) worn on each ankle during routine daily activities (e.g., cleaning, cooking, child care) to increase energy expenditure. The central hypothesis, based on existing literature and preliminary data, is that postpartum women with GDM will adopt an intervention that requires minimal additional time outside of their daily activities. We anticipate that this will result in additional weight loss that is clinically significant when compared with controls who only receive standard information on recommended physical activity. The rationale for the proposed research is that once an intervention that both improves T2DM factors and is easily adopted by women with GDM is known, early intervention specific to this restricted timeframe can be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Diagnosed with GDM in current pregnancy
* English language ability adequate for participation
* Plan to remain in the area for study duration
* Ability to provide informed consent

Exclusion Criteria:

* Prior Type 1 or Type 2 diabetes
* Pregnant with multiples (e.g., twin, triplets, etc.)
* Premature infant [<35 completed weeks gestation (assessed after delivery, before randomization)]
* Heart disease, serious illness, or conditions that may impede or prohibit participation in either study arm
* Pre-pregnancy BMI <18.5 (underweight)
* Live outside 35 mile radius of Ohio State University
* Woman is an appointed surrogate
* Infant will be adopted after delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We are assessing postpartum weight loss, therefore participants must be female to have the ability to give birth
Enrollment: 75 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Postpartum weight loss will be defined as weight change from initial weigh-in at NCH Visit 1 to final weigh-in at NCH Visit 2. Weight will be measured in person using the Tanita.

SECONDARY OUTCOMES:
Body Fat % | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Percent body fat will be defined as the change in initial measurement at NCH Visit 1 to final measurement at NCH Visit 2. Percent body fat will be measured in person using the Tanita.
BMI | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  BMI will be defined as the change from initial measurement at NCH Visit 1 to final measurement at NCH Visit 2. BMI will be measured using the Tanita for weight and obstetric medical record for height.
Waist-hip Ratio | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Waist circumference (cm) will be assessed at the middle point between the ribs and the iliac crest, with the participant standing. Hip circumference (cm) will be measured at the widest circumference of the buttocks. Change in circumference will be defined as the change from initial measurement at NCH Visit 1 to final measurement at NCH Visit 2. Waist-hip ratio will be measured in person using metric cloth tape.
Glycemia and Associated Biomarkers of Insulin Resistance and Metabolic Health: Oral Glucose Tolerance Test (OGTT) | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Blood will be collected during both visits at NCH and sent to the NCH lab for analysis. A fasting 2-hour, 75g OGTT will be conducted during both NCH visits. Glucose tolerance will be measured in mg/dL.
Glycemia and Associated Biomarkers of Insulin Resistance and Metabolic Health: HOMA | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Blood will be collected during both visits at NCH and sent to the NCH lab for analysis. Insulin sensitivity (β-cell function) will be measured using the Matsuda index and HOMA-IR. Matsuda index score and HOMA-IR will be determined based on insulin values (μU/mL) and glucose values (mg/dL) obtained from the OGTT.
Glycemia and Associated Biomarkers of Insulin Resistance and Metabolic Health: Hemoglobin A1c (HbA1c) | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Blood will be collected during both visits at NCH and sent to the NCH lab for analysis. HbA1c will be analyzed as a percentage.
Glycemia and Associated Biomarkers of Insulin Resistance and Metabolic Health: Leptin | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Blood will be collected during both visits at NCH and sent to the NCH lab for analysis. Fasting serum leptin will be measured in ng/mL.
Glycemia and Associated Biomarkers of Insulin Resistance and Metabolic Health: High sensitivity c-reactive protein (hs-CRP) | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Blood will be collected during both visits at NCH and sent to the NCH lab for analysis. hsCRP will be measured in mg/L.
Glycemia and Associated Biomarkers of Insulin Resistance and Metabolic Health: Adiponectin | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Blood will be collected during both visits at NCH and sent to the NCH lab for analysis. Adiponectin will be measured in µg/mL.
Glycemia and Associated Biomarkers of Insulin Resistance and Metabolic Health: Lipid Panel | NCH Visit 1 (25-35 days postpartum) to NCH Visit 2 (220-240 days postpartum)
  Blood will be collected during both visits at NCH and sent to the NCH lab for analysis. Lipids will be analyzed including total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and triglycerides. Lipids will be measured in mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Keim, PhD, MA, MS, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Racke CA, Keim SA, Yisahak SF, Stith BJ, Thung SF, Klebanoff MA, Gabbe SG, Landon MB, Oza-Frank R. Postpartum Physical Activity Intervention Among Women With Gestational Diabetes: A Randomized Controlled Trial. Am J Lifestyle Med. 2025 Jun 14:15598276251351809. doi: 10.1177/15598276251351809. Online ahead of print. PMID 40535905
- [Derived] Stith BJ, Buls SM, Keim SA, Thung SF, Klebanoff MA, Landon MB, Gabbe SG, Gandhi KK, Oza-Frank R. Moms in motion: weight loss intervention for postpartum mothers after gestational diabetes: a randomized controlled trial. BMC Pregnancy Childbirth. 2021 Jun 29;21(1):461. doi: 10.1186/s12884-021-03886-3. PMID 34187391